CLINICAL TRIAL: NCT05293223
Title: An Open-label Clinical Trial Phase IIB to Evaluate the Immunogenicity and Safety of Recombinant Novel Coronavirus Vaccine in Participants Aged 18 Years and Above That Previously Received One Dose of Sputnik V
Brief Title: Phase IIB Study of Recombinant Novel Coronavirus Vaccine
Acronym: FH-63
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: Dalhousie University (Other); CanSino Biologics Inc. (Industry)
Responsible Party: Principal Investigator, Pedro Cahn, PhD,Principal Investigator, Fundación Huésped
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FH-63 (CS-nCoV-SeqAD26)
Record Dates: First submitted 2021-11-24; First posted 2022-03-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: COVID-19 Vaccine
MeSH Terms: interventions — Ad5-nCoV vaccine

STUDY DESIGN:
Intervention Model Description: The ratio of Geometric mean titers (GMTs) of SARS-CoV-2 neutralizing antibody in participants on Day 21 post-vaccination of Ad5-nCoV (previously received a 1st dose of Sputnik V) (Group A) and two doses of Sputnik V (Group B) is used for the evaluation of this hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): One dose Sputnik V + one dose Ad5-nCoV
  Interventions: Biological: Ad5-nCov
- Group B (No Intervention): Samples stored at the immunology lab of the Buenos Aires University Medical School, corresponding to individuals vaccinated with 2 doses of Sputnik V.

INTERVENTIONS:
Biological: Ad5-nCov — Participants enrolled in Group A with only the 1st dose of Sputnik V will receive Ad5-nCoV vaccine at least 21 days but no more than 180 days after the first dose. They will be followed to evaluate the immunogenicity and safety of Ad5-nCoV vaccine during 6 months
  Arms: Group A

SUMMARY:
This is an open-label and non-randomized study to demonstrate the immunogenicity and safety profile in adults that received the Ad5-nCoV vaccine at least 21 days but no later than 90 days after the first dose of Sputnik V.

The non-inferiority hypothesis is used for the evaluation of the exploratory objective. The ratio of Geometric mean titers (GMTs) of SARS-CoV-2 neutralizing antibody in participants on Day 21 post-vaccination of Ad5-nCoV (previously received a 1st dose of Sputnik V) (Group A) and two doses of Sputnik V (Group B) is used for the evaluation of this hypothesis.

It is assumed to enroll about 100 subjects for each group. Additionally, 45 participants will be selected from Group A (to enter the immunogenicity subgroup for cellular immune response analysis. According to the above, considering extra subjects for compensating about 10% dropouts, the sample size of Group A is designed to be 450, for Group B is 200. Participants enrolled in Group A (1st dose of Sputnik V plus 1 dose of Ad5-nCoV) must have only received the 1st dose of Sputnik V and the interval between the previous injection (1st dose of Sputnik V) and the day of vaccination with Ad5-nCoV should be between 21 and 90 days. The comparator (Group B) will be the samples stored at the immunology lab of the Buenos Aires University Medical School, corresponding to individuals vaccinated with 2 doses of Sputnik V.

UPDATE : It's worth noting that enrollment number during the study was lower than the originallyplanned. According to the Protocol Group A sample size was designed to be 450. A low enrollment rate due to a fast vaccination rate (second dose) through the national COVID vaccination campaign for the entire population of Argentina resulted in difficulties in reaching the sample size planned. (the final number of participants enrolled and vaccinated in the study was 86 in arm A ).The enrollment period was affected due to the fast expansion of the National Vaccination Plan and the opportunity for potential participants to access it. Therefore, it was not possible to achieve the number of enrolled participants that was planned at the beginning of the study (450).

DETAILED DESCRIPTION:
There are 4 planned site visits in total: V1 (day0), V2 (day21), V3 (month 3), V4 (month 6) Healthy adults aged 18 years and above in Argentina will be informed by a procedure approved by the ethical review committee before consent is sought to be a volunteer. After passing the physical examination and screening according to the inclusion and exclusion criteria, they will be eligible to participate in this study.

Group B is a comparator group, in which samples stored corresponding to individuals who have already received 2 doses of Sputnik V will be used for the immunogenicity evaluation.

Study Procedures

* Informed consent
* Check inclusion and exclusion criteria All inclusion and exclusion criteria will be checked at the screening in-person visit and be reviewed at each in-person visit.
* Collect demographic data and contact information
* Medical history Obtain the participant's medical history by interview and/or review of the participant's medical records and record any pre-existing conditions or signs and/or symptoms present prior to injection in the EDC. This will include reviewing of any health condition that may prevent the participant from enrolling in the study, such as an unstable health condition or known positive HIV status (with less than 200 CD4 cells/mL).
* Check contraindications, warnings and precautions to injection Contraindications, warnings and precautions to injection must be checked before vaccination.
* Urine Pregnancy Test/Birth Control Women of child-bearing age will be asked to perform a urine pregnancy test at the day of enrollment. The result of the urine pregnancy test must be negative. In addition, participants who are able to become pregnant or could impregnate a partner are required to have used approved contraception at least 30 days prior to the study vaccination and for 90 days' post-vaccination.
* Physical examination Screening conclusion Participants will be deemed eligible to participate upon reviewing medical history and inclusion and exclusion criteria. This will occur prior to vaccination.
* Study group and treatment number allocation The eligible participants will be enrolled into Group A. Each participant will be assigned a treatment identification number (Subject ID).
* Check and record prior medications and concomitant medication/injection
* Check and record intercurrent medical conditions
* Pre-vaccination serology Approximately 10 mL of whole blood will be collected from each participant in Group A at Day 0 and separated for serum.
* Injection of study vaccine After completing all prerequisite procedures prior to injection, one dose of the assigned vaccine will be administered IM in the deltoid muscle of the upper arm for participants in Group A.
* Safety participant contacts Participants in group A need to record any AEs they may experience within 21 days post-vaccination. There is an on-site visit on the 21st day post-vaccination and the subjects need to submit their diary card.

Following up serology All participants in group A will have an in-person visit at Day 21, Month 3, and Month 6 post-vaccination of either Ad5-nCoV. Approximately 10 mL of whole blood will be collected from each participant and separated for serum.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years and above at the time of randomization.
2. Provide written informed consent.
3. Axillary temperature ≤ 37℃.
4. Never received any investigational or licensed COVID-19 vaccine other than the 1st dose of Sputnik V with an interval of 21-90 days before the study.
5. Subjects are eligible for immunization of this product as evaluated by investigators after medical history examination, physical examination and clinical judgment of health.

Exclusion Criteria:

1. Have a history of seizures, epilepsy, encephalopathy, psychosis.
2. History of anaphylaxis to any vaccine component.
3. Positive urine pregnancy test result, pregnant, lactation women, or intend to become pregnant within the next 6 months.
4. Congenital or acquired angioedema/neuroedema.
5. Medical history of Guillain-Barré syndrome.
6. Asplenia or functional absence of spleen.
7. Bleeding disorder (e.g. protein S or factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
8. Any confirmed or suspected immunosuppressive or immunodeficient state; received immunosuppressive therapy, cytotoxic therapy, or chronic corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis) within the past 6 months,
9. History of chronic systematic infection.
10. Administration of immunoglobulins and/or any blood products within three months prior to the planned administration of the vaccine candidate.
11. Receiving anti-tuberculosis or cancer treatment.
12. History of laboratory-confirmed COVID-19, or has a positive result at the examination of SARS-CoV-2 antigen before vaccination.
13. Planned to receive any vaccine (licensed or investigational), other than the study intervention, within 14 days before and after study vaccination.
14. Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e. warfarin) or novel oral anticoagulants (i.e. apixaban, rivaroxaban, dabigatran and edoxaban).
15. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, and affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The Geometric mean titers (GMTs) of SARS-CoV-2 neutralizing antibody | 21 days from baseline
  The Geometric mean titers (GMTs) of SARS-CoV-2 neutralizing antibody on Day 21 post-vaccination of Ad5-nCoV.

SECONDARY OUTCOMES:
The Geometric mean titers (GMTs) of SARS-CoV-2 neutralizing antibody | Month 3 and Month 6 from baseline
  The GMT of SARS-CoV-2 neutralizing antibody on Month 3 and Month 6 post-vaccination of Ad5-nCoV or the 2nd dose of Sputnik V.
solicited adverse events | from baseline to 7 days post-vaccination
  The incidence of solicited adverse reactions (ARs) within 7 days post-vaccination of Ad5-nCoV.
SARS-CoV-2 specific T-cell response | Day 21 post-vaccination of Ad5-nCoV
  The SARS-CoV-2 specific T-cell response is studied using flow cytometry, evaluating the expression of activation markers in T CD4+ and CD8+ cells. Expression of CD40L (CD154), and the production of interferon γ (IFN-γ), interleukin-2 (IL-2) and tumoral necrosis factor (TNF-α) will be studied.
The GMT of S-protein receptor binding domain (S-RBD) antibody | Day 21, Month 3, and Month 6
  The GMT of S-protein receptor binding domain (S-RBD) antibody on Day 21, Month 3, and Month 6 post-vaccination of Ad5-nCoV or the 2nd dose of Sputnik V.
unsolicited adverse events (AEs) | from baseline to 21 days post-vaccination
  To evaluate the incidence of unsolicited adverse events (AEs) within 21 days post-vaccination of Ad5-nCoV.
serious adverse events (SAEs) | from baseline to week 24
  The incidence of serious adverse events (SAEs) within 6 months post-vaccination of Ad5-nCoV.

CONTACTS AND LOCATIONS:
Locations (3):
- Argentina (3):
  - Fundación Huésped, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Centro de vacunación PREVIVAX, Ciudad Autonoma de Buenos Aire, Ciudad Autónoam de Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular CIPREC, Buenos Aires

DOCUMENTS (1):
  • Study Protocol (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT05293223/Prot_000.pdf